CLINICAL TRIAL: NCT00408434
Title: A Phase I Dose Finding Study of an Experimental New Drug, PPARγ Agonist Taken by Mouth by Patients With Advanced or Malignancies
Brief Title: Study of an Experimental New Drug, PPARγ Agonist Taken by Mouth by Participants With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-U102
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Neoplasm
Keywords: PPARγ agonist; advanced or metastatic malignancies; Tumor; Cancer
MeSH Terms: conditions — Neoplasms | interventions — efatutazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-7017 (Experimental): CS-7017 from 0.05 to 3.2 mg bid
  Interventions: Drug: CS-7017

INTERVENTIONS:
Drug: CS-7017 — CS-7017 0.05mg and 1.0mg tablets

SUMMARY:
An open-label, Phase I, dose escalation study of CS-7017 administered by mouth in sequential cohorts of 3 to 6 participants with advanced or metastatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed advanced or metastatic malignancy that is refractory to, not curable with, or not eligible for standard treatment(s).
* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Resolution of any toxic effects of prior therapy (except alopecia) to National Cancer Institute Common Terminology Criteria for Adverse Events v3.0 grade less than or equal to 1.
* Adequate organ and bone marrow function.
* Willing to use effective contraceptive while on treatment through at least 3 months thereafter.
* Negative pregnancy test for females of childbearing potential.
* Echocardiogram with ejection fraction within normal range.

Exclusion Criteria:

* Anticipation of need for a major surgical procedure or radiation therapy during the study.
* Treatment with chemotherapy, hormonal therapy, other thiazolidinediones, radiotherapy, minor surgery, or any investigational agent within 4 weeks (6 weeks for nitrosoureas, mitomycin C, immunotherapy, biological therapy, or major surgery) of study treatment start.
* Participants with clinically significant pleural or pericardial effusion (participants with minimal pleural effusion may be eligible at the Investigator's discretion).
* Clinically significant active infection, which requires antibiotic therapy, or human immunodeficiency virus (HIV)-positive participants receiving antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Clinical Lead, Study Director — Daiichi Sankyo
Locations (2):
- United States (2):
  - Washington D.C., District of Columbia
  - Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Pishvaian MJ, Marshall JL, Wagner AJ, Hwang JJ, Malik S, Cotarla I, Deeken JF, He AR, Daniel H, Halim AB, Zahir H, Copigneaux C, Liu K, Beckman RA, Demetri GD. A phase 1 study of efatutazone, an oral peroxisome proliferator-activated receptor gamma agonist, administered to patients with advanced malignancies. Cancer. 2012 Nov 1;118(21):5403-13. doi: 10.1002/cncr.27526. Epub 2012 May 8. PMID 22570147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants who met all inclusion criteria and no exclusion criteria were enrolled in study from 20 November 2006 to 03 April 2009 at 2 clinic sites in the United States. Of the 32 participants enrolled, 31 participants were dosed and received treatment.
Pre-assignment Details: Participants received CS-7017 (0.10 mg to 1.15 mg) every 12 hours. At least 3 participants were treated at each dose level. Dose escalation occurred after at least 3 participants in the current dosing cohort completed 1 cycle of treatment (3 weeks).
Groups:
- CS-7017 0.10 mg: Participants who received oral CS-7017 0.10 mg every 12 hours.
- CS-7017 0.15 mg: Participants who received oral CS-7017 0.15 mg every 12 hours.
- CS-7017 0.25 mg: Participants who received oral CS-7017 0.25 mg every 12 hours.
- CS-7017 0.35 mg: Participants who received oral CS-7017 0.35 mg every 12 hours.
- CS-7017 0.50 mg: Participants who received oral CS-7017 0.50 mg every 12 hours.
- CS-7017 0.75 mg: Participants who received oral CS-7017 0.75 mg every 12 hours.
- CS-7017 1.15 mg: Participants who received oral CS-7017 1.15 mg every 12 hours.
Period: Overall Study
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg
Started | 6 | 3 | 6 | 3 | 6 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 6 | 3 | 6 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 6 | 3 | 4 | 3 | 3 | 1 | 4
Not completed — Other | 0 | 0 | 1 | 0 | 2 | 1 | 0
Not completed — Terminated by Investigator | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg | Total
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 4 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.2) | 57.0 (14.7) | 58.7 (8.8) | 58.7 (13.7) | 62.3 (8.6) | 52.3 (11.1) | 53.5 (7.6) | 58.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 4 | 0 | 2 | 0 | 0 | 9
  Male | 3 | 3 | 2 | 3 | 4 | 3 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 3 | 6 | 1 | 6 | 3 | 4 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 6 | 3 | 6 | 3 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response Following Administration of CS-7017 in Participants With Advanced or Metastatic Malignancies
Description: Complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions). Objective response rate was defined as the sum of all CRs and PRs.
Time Frame: Baseline up to at least 2 cycles (each cycle was 3 weeks), up to 2 years 5 months
Population: Best overall response was assessed in the Efficacy Population.
Measure: Count of Participants; unit: Participants
Groups:
- CS-7017 All Participants: All participants who received CS-7017 with doses ranging from 0.10 mg to 1.15 mg every 12 hours.
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg | CS-7017 All Participants
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 5 | 3 | 3 | 27
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Stable disease (SD) | 3 | 2 | 0 | 1 | 4 | 1 | 1 | 12
  Progressive disease (PD) | 3 | 1 | 4 | 2 | 1 | 1 | 2 | 14
  Objective response rate (CR+PR) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

2. Secondary Outcome: Summary of Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve of Means of Serum Free Form of CS-7017 (R-150033) Following Administration of CS-7017 in Participants With Advanced or Metastatic Malignancies
Description: Area under the plasma/serum drug concentration-time curve for dosing interval (AUC[0-tau]), computed using the linear trapezoidal rule and area under the plasma/serum drug concentration-time curve from 0 to last time point above the quantification limit (AUC[0-t]) calculated using the linear trapezoidal rule were assessed.
Time Frame: Day 1 of Cycles 1 and 2: predose, 0.5, 1, 2, 3, 4, 6, and 10 hours postdose; and predose on Day 8 and 15 of Cycle 1.
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 4
ng*h/ml
  AUC(0-tau) | 23.05 (6.11) | 32.05 (7.75) | 68.33 (24.61) | 59.72 (32.58) | 159.2 (45.10) | 159.14 (126.31) | 256.3 (93.31)
  AUC(0-12): number analyzed (Participants) | 5 | 3 | 6 | 3 | 6 | 3 | 4
  AUC(0-12) | 32.96 (6.90) | 44.14 (12.15) | 91.24 (36.16) | 80.80 (40.74) | 220.9 (74.42) | 214.38 (163.81) | 356.8 (127.69)

3. Secondary Outcome: Summary of Pharmacokinetic Parameter Observed Maximum Plasma Concentration (Cmax) of Means of Serum Free Form of CS-7017 (R-150033) Following Administration of CS-7017 in Patients With Advanced or Metastatic Malignancies
Description: Cmax was defined as observed maximum plasma concentration.
Time Frame: Day 1 of Cycles 1 and 2: predose, 0.5, 1, 2, 3, 4, 6, and 10 hours postdose; and predose on Day 8 and 15 of Cycle 1.
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 4
ng/ml | 4.21 (0.93) | 5.76 (1.53) | 12.19 (3.00) | 12.26 (7.10) | 26.92 (6.36) | 27.64 (21.44) | 44.73 (15.05)

4. Secondary Outcome: Summary of Pharmacokinetic Parameter Terminal Elimination Half-life (t1/2) of Means of Serum Free Form of CS-7017 (R-150033) Following Administration of CS-7017 in Patients With Advanced or Metastatic Malignancies
Time Frame: Day 1 of Cycles 1 and 2: predose, 0.5, 1, 2, 3, 4, 6, and 10 hours postdose; and predose on Day 8 and 15 of Cycle 1.
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 4
hour | 8.51 (3.92) | 13.78 (6.92) | 11.48 (11.30) | 12.49 (7.35) | 5.74 (2.56) | 9.08 (2.79) | 11.66 (3.45)

5. Secondary Outcome: Summary of Pharmacokinetic Parameter Time of Maximum Plasma Concentration (Tmax) of Means of Serum Free Form of CS-7017 (R-150033) Following Administration of CS-7017 in Patients With Advanced or Metastatic Malignancies
Description: Tmax was defined as time of maximum plasma concentration.
Time Frame: Day 1 of Cycles 1 and 2: predose, 0.5, 1, 2, 3, 4, 6, and 10 hours postdose; and predose on Day 8 and 15 of Cycle 1.
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Population.
Measure: Mean (Full Range); unit: hour
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 4
hour | 3.00 [2.00 to 6.00] | 2.00 [1.00 to 2.00] | 1.58 [1.00 to 4.00] | 3.00 [1.00 to 3.00] | 2.00 [1.00 to 4.00] | 3.00 [2.00 to 4.00] | 2.50 [2.00 to 4.00]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) data were collected from baseline up to 30 days after the last dose of study drug, up to 2 years 5 months.
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the first dose until 30 days after the last dose.
Arm/Group | CS-7017 0.10 mg | CS-7017 0.15 mg | CS-7017 0.25 mg | CS-7017 0.35 mg | CS-7017 0.50 mg | CS-7017 0.75 mg | CS-7017 1.15 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 2/3 | 0/6 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/3 | 2/6 | 2/3 | 3/6 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/6 | 3/3 | 6/6 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.10 mg (N=6) | CS-7017 0.15 mg (N=3) | CS-7017 0.25 mg (N=6) | CS-7017 0.35 mg (N=3) | CS-7017 0.50 mg (N=6) | CS-7017 0.75 mg (N=3) | CS-7017 1.15 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overloading (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.10 mg (N=6) | CS-7017 0.15 mg (N=3) | CS-7017 0.25 mg (N=6) | CS-7017 0.35 mg (N=3) | CS-7017 0.50 mg (N=6) | CS-7017 0.75 mg (N=3) | CS-7017 1.15 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 6 | 1 | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 4 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 3 | 1 | 6 | 2 | 4
Oedema peripheral (General disorders) | 6 | 1 | 3 | 1 | 3 | 2 | 1
Weight increased (Investigations) | 5 | 2 | 4 | 1 | 1 | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 3 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 2 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No